CLINICAL TRIAL: NCT05492383
Title: SAvvyWire™ EFficacy and SafEty in Transcatheter Aortic Valve Implantation Procedures (SAFE-TAVI)
Acronym: SAFE-TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Opsens, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRT-2015-32
Record Dates: First submitted 2022-07-26; First posted 2022-08-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Severe Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized, single-arm, multicenter, clinical performance pivotal clinical investigation.
Masking Description: Investigation participant number only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with severe symptomatic AS undergoing TAVI (Experimental): Patients with severe symptomatic AS undergoing a TAVI procedure with a THV for which rapid pacing is considered necessary during valve implantation
  Interventions: Device: TAVI

INTERVENTIONS:
Device: TAVI — Patients with severe symptomatic AS undergoing Transcatheter aortic valve implantation (TAVI)

SUMMARY:
The purpose of the clinical investigation is to determine efficacy and safety of using the rapid pacing of SavvyWire™ during TAVI procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject has a severe symptomatic AS undergoing a TAVI procedure
3. Subject with a THV for which rapid pacing is considered necessary during valve implantation
4. Subject agrees to participate in the study and is able to sign the informed consent form

Exclusion Criteria:

1. Failure to provide signed informed consent
2. Extremely horizontal aorta (aortic root angle ≥70°)
3. Extreme tortuosity at the level of the iliofemoral arteries, thoracic or abdominal aorta
4. Inability to receive full anticoagulation during the TAVI procedure
5. Prohibitive surgical risk precluding (according to the Heart Team) conversion to open heart surgery in case of a life-threatening complication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with effective rapid pacing run | during surgery
  Effective rapid pacing will be defined as an adequate ventricular pacing capture by the SavvyWireTM leading to a reduction of systolic aortic pressure value <60 mmHg.

SECONDARY OUTCOMES:
Presence of major complications (safety) | during surgery
  Presence of major complications related to the SAVVY guidewire including guidewire kink hindering or preventing the advancement of the transcatheter valve system, left ventricular perforation and pacing capture translating into major clinical consequences (transcatheter valve malpositioning or embolization).
Percentage of patients with hemodynamic assessment without additional manipulation (pressure efficacy) | during surgery
  Ventricular pressure recording with the SavvyWireTM, allowing gradient calculation and display by the OptoMonitor 3, without the need of additional device exchanges through the aortic valve after valve implantation.
Percentage of patient with valve advancement to intended position (mechanical efficacy) | during surgery
  Effective advancement of the THV delivery system over the SavvyWireTM allowing a precise positioning of the valve to the intended deployment position.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodés-Cabau, Dr, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (6):
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Álvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Regueiro A, Alperi A, Vilalta V, Asmarats L, Baz JA, Nombela-Franco L, Calabuig A, Munoz-Garcia A, Sabate M, Moris C, Picard-Deland M, Pelletier-Beaumont E, Rodes-Cabau J. Safety and Efficacy of TAVR With a Pressure Sensor and Pacing Guidewire: SAFE-TAVI Trial. JACC Cardiovasc Interv. 2023 Dec 25;16(24):3016-3023. doi: 10.1016/j.jcin.2023.10.035. Epub 2023 Oct 23. PMID 37902144